CLINICAL TRIAL: NCT01311947
Title: Relation of Hepatitis B Virus Mutants and the Therapeutic Effect of Peginterferon Alfa-2a in HBeAg-Positive Chronic Hepatitis B
Brief Title: Hepatitis B Virus Mutants and the Therapeutic Effect of Peginterferon Alfa-2a in HBeAg-Positive Chronic Hepatitis B
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Cheng-Yuan Peng, Director of Division of Hepatogastreoenterology, China Medical University Hospital
Other Study IDs: DMR99-IRB-313
Record Dates: First submitted 2011-03-08; First posted 2011-03-10 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Hepatitis B, Chronic
Keywords: Chronic hepatitis B; Peginterferon alfa-2a
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Serum specimens
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Peginterferon alfa-2a — Peginterferon alfa-2a at 180 ug weekly for 24 weeks
  Other Names: Pegasys

SUMMARY:
In order to clarify the association between HBV mutations appearing before and during interferon therapy and the therapeutic effects, serial serum samples from 100 HBeAg-positive CHB patients undergoing peginterferon alfa-2a therapy will be collected and analyzed for the mutations of preS/S gene and BCP-preC/C region, particularly for the deletion mutations. Furthermore, Real-Time PCR will be performed to measure the ratios of wild-type HBV and deletion mutant HBV before and at the end of peginterferon alfa-2a therapy. Finally, statistical analysis will be done to elucidate whether the mutations of preS/S gene and BCP-preC/C region have any relation with the therapeutic effect of peginterferon alfa-2a.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) infection is a serious worldwide health issue. Approximately 400 million people worldwide are chronic hepatitis B (CHB) patients. Currently, two therapeutic methods can be used to treat CHB. One is the nucleos(t)ide analogues, the other is the interferon alfa. Interferon alfa acts mainly by enhancing the immune system and directly inhibits the virus to a limited extent. It is known that mutations at preS, S, basal core promoter, precore and core gene are associated with an increased risk of HCC. However, it remains to be clarified as to the relation between HBV mutations and the therapeutic responses to interferon treatment. In order to clarify the association between HBV mutations appearing before and during interferon therapy and the therapeutic effects, serial serum samples from 100 HBeAg-positive CHB patients undergoing peginterferon alfa-2a therapy will be collected and analyzed for the mutations of preS/S gene and BCP-preC/C region, particularly for the deletion mutations. Furthermore, Real-Time PCR will be performed to measure the ratios of wild-type HBV and deletion mutant HBV before and at the end of peginterferon alfa-2a therapy. Finally, statistical analysis will be done to elucidate whether the mutations of preS/S gene and BCP-preC/C region have any relation with the therapeutic effect of peginterferon alfa-2a.

ELIGIBILITY:
Inclusion Criteria:

HBeAg-positive chronic hepatitis B patients on Peginterferon therapy

Exclusion Criteria:

HBeAg-negative chronic hepatitis B patients HBeAg-positive chronic hepatitis B patients on other kinds of therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HBeAg-positive chronic hepatitis B
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Therapeutic response to Peginterferon Alfa-2a in HBeAg-Positive Chronic Hepatitis B | 24 weeks after the end of 24 weeks of Peginterferon alfa-2a treatment

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Yuan Peng, MD, PhD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan, Taiwan

REFERENCES:
- [Background] Desmond CP, Bartholomeusz A, Gaudieri S, Revill PA, Lewin SR. A systematic review of T-cell epitopes in hepatitis B virus: identification, genotypic variation and relevance to antiviral therapeutics. Antivir Ther. 2008;13(2):161-75. PMID 18505168